CLINICAL TRIAL: NCT05500105
Title: Remote Delivery of a Visuospatial Intervention, Involving Tetris Computer Game Play, to Reduce Intrusive Memories in Parents After Paediatric Intensive Care Intensive Care: a Feasibility Study
Brief Title: Remote Delivery of a Visuospatial Intervention to Reduce Traumatic Intrusive Memories After Paediatric Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, David McCormack, Clinical Director, Doctorate in Clinical Psychology Programme, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPS 22_57
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Intrusion Symptom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simple cognitive task intervention (Experimental): Session 1: A memory cue followed by playing the computer game "Tetris" (e.g. on own smartphone) with mental rotation instructions.
  Options to engage in self-administered/guided booster sessions per intrusive memory.
  Interventions: Other: Simple cognitive task intervention

INTERVENTIONS:
Other: Simple cognitive task intervention — Session 1: A memory cue followed by playing the computer game "Tetris" (e.g. on own smartphone) with mental rotation instructions.
  Options to engage in self-administered/guided booster sessions per intrusive memory.

SUMMARY:
This study aims to examine the feasibility and acceptability of a brief intervention, involving a imagery-competing task, remotely delivered to parents who are currently experiencing persistent intrusive traumatic memories at least one month following their child's discharge from intensive care.

DETAILED DESCRIPTION:
This is a feasibility study of a brief intervention, involving a visuospatial intervention (i.e. an imagery-competing task), remotely delivered to parents who are currently experiencing persistent intrusive traumatic memories at least one month following their child's discharge from the paediatric intensive care unit (PICU) or neonatal intensive care (NICU).

This study seeks to examine the feasibility and acceptability of delivering this brief intervention remotely with parents currently experiencing persistent intrusive traumatic memories at least one month following their child's discharge from PICU or NICU. The study aims to estimate recruitment, retention, outcome completion and adherence rates, assess acceptability, and in addition to explore the preliminary effect of the intervention on primary and secondary outcomes. Specifically, this study seeks to answer the following questions:

1. How willing are parents, who are currently experiencing persistent intrusive traumatic memories, at least one month following their child's discharge from PICU or NICU, to take part in this brief intervention delivered remotely?
2. How willing are parents to remain in the study until completion at follow up?
3. How willing are participants to complete all outcome measures?
4. How acceptable is this intervention to parents when delivered remotely?
5. Having taken part in the study, how willing are these parents to give consent for their child to take part in this intervention?
6. Having completed the intervention, how willing are parents to be part of a randomised control group?
7. Does this intervention help reduce the number of intrusive memories participants experience, as well as symptoms of anxiety, depression and PTS from baseline to follow-up?

Please note: After approximately six months into recruitment the enrolment target of 20 participants had not been achieved, only 12 participants had consented to take part in the study by this time. After reflecting on the recruitment process it was decided to include parents whose child had either been admitted to paediatric intensive care (PICU) or neonatal intensive care (NICU). The rationale for this was that research evidence demonstrates that admission to either a NICU or a PICU is similarly stressful for parents (Seideman et al., 1997) and many commonalities exist between them, "most notably the similarity of parent and staff experiences and the coexisting medical, psychological and developmental needs of babies and children" (Atkins & Syed-Sabir, 2022, p.9). Parents who have had a child in intensive care can experience intrusive memories whether that be paediatric or neonatal intensive care. Therefore, in light of this, it seemed worthwhile to see if explicitly seeking to recruit parents whose child had been admitted to PICU or NICU would improve participant enrolment. On 10th March 2023, after receiving approval from the research ethics committee, the study documents were amended (e.g., advert, participant information sheet etc.) to explicitly extend to parents who have had a child in intensive care to include parents whose child has been in either PICU or NICU.

ELIGIBILITY:
Inclusion Criteria:

1. Parent of a child who was discharged from PICU or NICU at least one month prior to study recruitment.
2. Parent who is currently experiencing persistent intrusive memories (at least a minimum of three intrusive memories in the past week).
3. Parent who has access to, and sufficient ability to use an electronic device (smartphone/tablet and/or computer/laptop) for remote delivery.
4. Adult aged 18 or older
5. Live in the UK or Ireland

Exclusion Criteria:

1. Parent of a child who was discharged from PICU or NICU less than one month prior to study recruitment.
2. Parent who experienced less than three intrusive memories in the past week
3. Parent who does not have access to, and ability to, use an electronic device e.g., computer or smartphone.
4. Younger than 18 years old
5. Does not live in the UK or Ireland

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event(s) - change in number of intrusive memories is being assessed. | At baseline for 7 days, After session 1 for 7 days, and 7 days prior to follow-up at one month post intervention.
  Number of intrusive memories of traumatic event(s) recorded by participants in a brief diary daily for 7 days.

SECONDARY OUTCOMES:
Impact of Events Scale-Revised (IES-R; Weiss and Marmar, 1997) | Baseline, 1 week follow-up, and 1 month follow-up
  Self-report measure that assesses subjective distress after a traumatic event (with reference to study event[s]) in the last week. Here we include the intrusion subscale (8 items) and the avoidance subscale (8 items). Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Subscale scores are calculated for the Intrusion or Avoidance items summed (ranging from 0 to 32 each). Higher scores indicate worse outcome.
Intrusive memory ratings | 1 week follow-up and 1 month follow-up
  It is a 9-item a self-report questionnaire which assesses a number of intrusive memories characteristics. It is adapted from an ongoing trial of the intervention in the UK (GAINS study; ClinicalTrials.gov Identifier: NCT04992390)
Patient Health Questionnaire-9 item (PHQ-9; Kroenke et al., 2001) | Baseline, 1 week follow-up, and 1 month follow-up
  It is a 9-item self-report measure of depressive symptoms.
Generalised Anxiety Disorder-7 item questionnaire (GAD-7; Spitzer et al., 2006) | Baseline, 1 week follow-up, and 1 month follow-up
  It is a 7-item self-report measure of generalised anxiety symptoms.
Work and Social Adjustment Scale (WSAS; Mundt et al., 2002) | Baseline, 1 week follow-up and 1 month follow-up
  It is is a 5-item scale measuring an individual's ability to function in five domains of everyday life; work, home management, social leisure activities, private leisure activities and close relationships.

OTHER OUTCOMES:
Self-administered use of the intervention | 1 week follow-up and 1 month follow-up
  It is a self-report measure containing 4 items which will be used to assess adherence to self-administered 'booster' sessions of the intervention. It is adapted from ongoing trial of the intervention in Sweden (EKUT-P study; ClinicalTrials.gov Identifier: NCT04460014)
Interview with participants regarding participation | 1 month follow-up
  A semi-structured interview regarding their experience of taking part in the study.

CONTACTS AND LOCATIONS:
Overall Officials: David McCormack, Dr, Principal Investigator — The Queen's University of Belfast; Lalitha Iyadurai, Dr, Principal Investigator — University of Oxford; Emily Holmes, Professor, Principal Investigator — Uppsala University / Karolinska Institutet
Locations (1):
- Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be made available starting 6 months after publication. An anonymised database of individual participant data, along with a data dictionary, as well as the Clinical Study Report (which will include summarised anonymised participant data), will be shared on the Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of a paper.
Access Criteria: All IPD that underlie results in a publication will be made available starting 6 months after publication. An anonymised database of individual participant data, along with a data dictionary, as well as the Clinical Study Report (which will include summarised anonymised participant data), will be shared on the Open Science Framework.